CLINICAL TRIAL: NCT05219825
Title: Breathwork-assisted Treatment for Cannabis Use Disorder: a Proof-of-concept Study
Brief Title: Breathwork-assisted Treatment for Cannabis Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elias Dakwar (Other)
Responsible Party: Sponsor-Investigator, Elias Dakwar, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8165
Record Dates: First submitted 2021-12-30; First posted 2022-02-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Addiction; Substance Abuse; Cannabis Use Disorder; Cannabis Use; Cannabis Dependence; Cannabis Abuse
Keywords: Addiction; cannabis use disorder; Breathwork; Non-ordinary states of consciousness; Non-ordinary experiences; Contemplative practices; Altered states of consciousness; Cannabis
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breathwork group (Experimental): Treatment-seeking individuals with cannabis use disorder who will participate in the 1-week breathwork workshop.
  Interventions: Behavioral: Breathwork workshop

INTERVENTIONS:
Behavioral: Breathwork workshop — Participants will complete 1.5 hours of breathwork session in addition to a total of 6 hours of brief psychotherapeutic intervention in a span of 1 week. The therapy sessions will occur both before and after the breathing session.
  Other Names: Enhanced breathing session + Brief psychotherapeutic intervention

SUMMARY:
The purpose of this proof-of-concept study is to evaluate the safety, feasibility and acceptability of a breathwork workshop intervention in individuals with cannabis use disorder.

DETAILED DESCRIPTION:
This study will test a 1-week breathwork workshop for treatment-seeking adults with a diagnosis of cannabis use disorder. The intervention consists of an enhanced breathing session with evocative music to facilitate experiencing non-ordinary states of consciousness, in addition to brief therapeutic interventions based on Motivational Interviewing and Mindfulness-based Relapse Prevention (MBRP). The primary aim is to test the acceptability, feasibility and safety of enhanced breathwork in a therapeutic framework for cannabis use disorder. In addition, the investigators seek to understand the phenomenology of breathwork that may explain any change related to addictive behaviors, as well as biological changes that occur during the breathwork session through heart rate variability and electroencephalography.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for active cannabis use disorder.
* Seeking treatment for their cannabis use

Exclusion Criteria:

* Meets DSM-V criteria for schizophrenia or any psychotic illness or any dissociative disorder (Dissociative identity disorder, Dissociative amnesia, Depersonalization/derealization disorder).
* Active substance use disorder except for cannabis, nicotine, and caffeine.
* History of severe withdrawal symptoms (i.e withdrawal seizures).
* History of dementia, epilepsy or seizures, cardiac arrhythmia, pacemaker/defibrillator, heart failure, asthma, panic disorder and other respiratory illnesses (ie: COPD).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the breathwork session | One week after the breathing session.
  Acceptability of the breathwork intervention through self-reported questionnaires.
Safety of the breathing session | 24 hours after the breathing session.
  Occurrence of adverse effects through a self-reported questionnaire.

SECONDARY OUTCOMES:
Change in Cue Reactivity | From baseline to 1 month after the breathing session.
  Serial visual analogue scale for craving elicited by cannabis use.
Change in Motivation to Quit | From baseline to 1 month after the breathing session.
  Measured with the "Stages of Change Readiness and Treatment Eagerness Scale."
Change in cannabis use | From baseline to 1 month after the breathing session.
  Changes in cannabis use as measured by the Timeline Followback.
Phenomenology of breathwork #1 | 24 hours after the breathing session
  Subjective experiences during the breathing session will be assessed with the 30-item Mystical Experience Questionnaire.
Phenomenology of breathwork #2 | Obtained 24 hours after the breathing session
  Subjective experiences during the breathing session will be assessed with the Emotional Breakthrough Inventory.
Heart Rate Variability | Measured during breathing session
  Polar (H10) chest strap
Electroencephalographic changes | Measured during breathing session
  Electroencephalograpy cap

CONTACTS AND LOCATIONS:
Overall Officials: Silvia J Franco Corso, M.D, Principal Investigator — New York State Psychiatric Institute/ Columbia University Medical Center; Elias Dakwar, M.D, Study Chair — New York State Psychiatric Institute/ Columbia University Medical Center; Kate O'Malley, M.A, Study Director — New York State Psychiatric Institute/ Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No